CLINICAL TRIAL: NCT02540707
Title: Comparisons of the Effects of Solifenacin Versus Mirabegron on Autonomic System, Arterial Stiffness and Psychosomatic Distress and Clinical Outcomes: A Prospective Randomized Controlled Trial
Brief Title: Comparisons of the Effects of Solifenacin Versus Mirabegron on Autonomic System, Arterial Stiffness and Psychosomatic Distress and Clinical Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201506092MIND
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solifenacin (Placebo Comparator): Women with overactive bladder syndrome will be treated by solifenacin 5 mg qd * 12 weeks
  Interventions: Drug: solifenacin
- Mirabegron (Experimental): Women with overactive bladder syndrome will be treated by mirabegron 25 mg qd * 12 weeks
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: solifenacin — solifenacin 5 mg per day for 12 weeks
  Arms: Solifenacin
Drug: mirabegron — mirabegron 25 mg per day for 12 weeks
  Arms: Mirabegron

SUMMARY:
Background/Purpose: The overactive bladder syndrome (OAB) affects around 17 % of female population. Antimuscarinics can affect autonomic system, arterial stiffness and psychosomatic distress. However, there is no such research for the new drug- mirabegron (a β3-agonist). Thus, the aim of our study is to analyze the between-group differences in heart rate variability, cardio-ankle vascular index, ankle-brachial pressure index, psychosomatic distress, personality trait, family support and clinical outcomes between the mirabegron and the solifenacin groups.

Patients and Methods: The investigators will perform a prospective randomized controlled study to recruit 150 female OAB patients at the outpatient clinic of Department of Obstetrics and Gynecology of National Taiwan University Hospital. All OAB female patients will be asked to complete Urgency Severity Scales, Overactive Bladder Symptoms Scores questionnaires, King's Health questionnaires, UDI-6 & IIQ-7, Patient Health Questionnaire, brief symptom rating scale (BSRS), Maudsley personality inventory (MPI) and adaptability, partnership, growth, affection, and resolve (APGAR) questionnaires, Sleep and Dietary habit Questionnaire, standard 12-leads electrocardiography (ECG), 5 minutes Holter monitoring, cardio-ankle vascular index (CAVI) test, bladder diary, 20-min pad test, urodynamic studies and measurement of urinary nerve growth factors level before and after 12 weeks' mirabegron versus solifenacin treatment. STATA software is used for statistical analyses.

Possible Results: The investigators can answer that the between-group differences in heart rate variability, cardio-ankle vascular index, ankle-brachial pressure index, psychosomatic distress, personality trait, family support and clinical outcomes between the mirabegron and the solifenacin groups. The above conclusions should be important for pre-treatment consultation.

ELIGIBILITY:
Inclusion Criteria:

* Women with overactive bladder syndrome
* ≥20 year-old

Exclusion Criteria:

* Urine retention,
* acute angle glaucoma,
* myasthenia gravis,
* ulcerative colitis,
* megacolon

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Between-group difference of the effect of drug on heart rate variability | 12 weeks
  Between-group difference of the effect of drug on heart rate variability, such as low frequency and high frequency
Between-group difference of the effect of drug on psychosomatic distress | 12 weeks
  Between-group difference of the effect of drug on psychosomatic distress by Brief Symptom Rating Scale

SECONDARY OUTCOMES:
Between-group difference of the effect of drug on arterial stiffness | 12 weeks
  Between-group difference of the effect of drug on arterial stiffness by cardio-ankle vascular index
Between-group difference of the effect of drug on clinical efficacy | 12 weeks
  Between-group difference of the effect of drug on clinical efficacy by Overactive Bladder Symptoms Score Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinics, Department of Obs/Gyn, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401